CLINICAL TRIAL: NCT03491930
Title: What is the Effect of a Feedback Device on Weight Loss and Metabolic Measurements in Obese People With the Metabolic Syndrome?
Brief Title: Weight Loss Using a Feedback Device in Obese People With the Metabolic Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never initiated. PI withdrew protocol with the IRB.
Sponsor: Rockefeller University (Other)
Collaborators: Molloy College (Other)
Responsible Party: Principal Investigator, Jeanne Walker, Clinical research nurse practitioner, Rockefeller University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JWA-0967
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Weight Loss; Obesity; Pre-Diabetes; Metabolic Syndrome
Keywords: Weight Loss; Obesity; Pre-Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Weight Loss; Obesity; Glucose Intolerance; Metabolic Syndrome | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A single group of participants will undergo study participation of listed interventions, over a 3 month outpatient period, to assess the effects on weight loss. A control group will receive all of the interactions and testing as the intervention group, except they will not use the weight loss app or receive weekly phone coaching.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Cohort (Experimental): VA MOVE! Coach app: Weight loss using the VA MOVE! Coach weight loss app which presents positive feedback, education in nutrition and portion sizes, coping mechanisms, charts and graphs. App will be used for three months.
  Telephone Coaching: Weekly phone coaching will provide further support and assist with problem solving and goal setting for a three month period.
  Standard of care for weight loss (the 2013 AHA/ACC/TOS guidelines). Followed for three months.
  Pre and post weight loss metabolic measurements will be obtained.
  Interventions: Device: VA MOVE! Coach app; Behavioral: Telephone Coaching; Behavioral: Standard of Care for weight loss.
- Control Cohort (Active Comparator): Standard of care for weight loss (2013 AHA/ACC/TOS guidelines). Followed for three months.
  Pre and post weight loss metabolic measurements will be obtained.
  Interventions: Behavioral: Standard of Care for weight loss.

INTERVENTIONS:
Device: VA MOVE! Coach app — The VA MOVE! Coach app promotes weight loss through positive feedback, nutritional education, calorie counts, graphs, charts, and encourages increased activity. Efforts will be supported through weekly phone coaching.
  Arms: Interventional Cohort
Behavioral: Telephone Coaching — Weekly Telephone Coaching
  Arms: Interventional Cohort
Behavioral: Standard of Care for weight loss. — Standard of Care for weight loss (2013 American College of Cardiology/American Heart Association Task Force and The Obesity Society (AHA/ACC/TOS) Report,PubMed Identification: 24222017).
  To include:
  * Vioscreen food frequency assessment and bionutritionist consult.
  * Healthy eating nutritional pamphlets (during consult)
  * Decrease daily caloric intake by 500 cal/day
  * Increase in physical activity (goal: 10,000 steps per day - measured by pedometer.)
  * Dietary counseling by Clinician (monthly)

SUMMARY:
The purpose of this study is to determine if a weight loss app (VA MOVE!® Coach App) along with regularly scheduled telephone counseling, will motivate obese people with metabolic syndrome to lose weight and improve the symptoms of the metabolic syndrome, compared to usual weight loss approaches. This study will randomly assign participants to one of two groups, interventional or control. The interventional group will use the app with phone coaching and standard of care for weight loss. The control group will receive standard weight loss care without the app and phone coaching. Weight loss motivation to adopt life-style changes to maintain weight loss and quality of life between the two groups will be compared. The metabolic syndrome (MetS) is a cluster of disorders including high blood pressure, pre-diabetes, the tendency to carry body weight around the waist, and increased fat in the blood. When these problems happen together, there is an increased risk for heart attack, stroke, diabetes and certain cancers.

Although the metabolic syndrome is a serious condition, it can be treated with diet, weight loss and increased activity. It can even be reversed using these lifestyle changes. Due to poor success with routine short-term weight loss treatment (group and one-on-one counseling), it is time to address the problem by a different method. Studies have shown feedback devices and weight loss apps have been successful in weight loss and weight maintenance. They are economical (many apps are free), and convenient to use, without attendance at group sessions. Since weight loss is the corner stone for improvement in the symptoms of the MetS, this study will offer a unique approach to support individuals who are committed to losing weight and adopting a healthier lifestyle.

Numerous studies demonstrated that feedback via text messaging, and interaction through social networking support groups, in addition to iPhone apps, are all more effective in weight loss measures than group sessions at a hospital site. (Duncan et al., 2011; Greene, Sacks, Piniewski, Kil, & Hahn, 2012; Shaw et al., 2013; Spring et al., 2013). The benefit of these various methods is that they appear to accelerate weight loss and prevent weight re-gain if employed long-term. With technology changing daily, these approaches must be considered an essential adjunct to, or replacement for, traditional group counselling sessions.

DETAILED DESCRIPTION:
Obesity rates in the United States have steadily increased since the 1980's, doubling between 1980 and 2010 from 15.0% to 36.1% (Cefalu et al., 2015). The prevalence rate of obesity in adults in the U.S. in 2014 was 37.7%, according to the Centers for Disease Control and Prevention (CDC) National Center for Health Statistics (Ogden, Carroll, Fryar, & Flegal, 2015) resulting in a rising incidence of type 2 diabetes, heart disease, hypertension, and some cancers (American Society of Clinical Oncology, 2014). Many contributors to the rise in obesity rates are cited in the literature: socio-economic, urbanization, sedentary behavior (Hruby & Hu, 2015), psychological and motivational factors (Byrne, Cooper, & Fairburn, 2003), and ethnicity and gender (Ogden et al., 2015). ). According to research done by The Pew Research Center (DeSilver, 2016), daily caloric intake by the average American in 2010 was 2,481 calories, about 23% more than in 1970.

As research into obesity continues, contributing factors include more than excessive dietary intake and decreased physical activity. Obesity scientists and medical specialists view the disorder as a systemic dynamic involving the brain, gut, liver, adipose tissue, hormones, inflammation, and heredity (Cefalu et al., 2015). The condition, recognized by the American Medical Association as a disease in 2011, resulted in obesity specialists and medical board certification (American Board of Obesity Medicine, ABOM, 2013).

Though considered a disease in itself, obesity is a major contributor to preventable morbidity and mortality, as well as to enormous health care costs (American Nurse Practitioner Foundation, 2013). The estimated cost of obesity and the resultant co-morbidities in the U.S. in 2015 was $190 billion. This figure represented 21% of total U.S. healthcare costs (Hruby & Hu, 2015). Furthermore, the excess cost incurred by obese individuals annually over the non-obese was $1,152 for obese men (for prescription drugs and hospitalizations), and $3,613 for obese women (Hruby & Hu, 2015).

Nearly 35% of all adults and 50% of those over 60 years of age in the United States, have the Metabolic Syndrome (MetS) (Aguilar et al 2015). This is especially disturbing since the population over 60 years of age increases annually, due to the aging of America. Obesity and the MetS are the underlying factors in most of the chronic illnesses prevalent today: diabetes, cancer, inflammatory diseases, reduced immunity, heart disease, stroke, and disability. It is clear that new, pragmatic, cost effective treatment to control the risk factors and resultant morbidity and mortality, caused by this epidemic, must be aggressively investigated. Employing apps developed for mobile phones is an obvious choice, if the data can show evidence that this approach is effective. This is a prime area for nurse practitioners to initiate research and to add to the scientific knowledge of obesity and its sequelae (American Nurse Practitioner Foundation, 2013).

This will be the first study of its kind to examine changes in the metabolic markers of the MetS, body composition and biometrics using a feedback device in the form of a weight loss app. As such, it has the potential to provide clinicians with evidence based, adjunctive treatment for this population. This study will provide the seeds for a longer study to determine the feasibility of using feedback devices to reinforce healthy life styles and continue or maintain the weight loss. In this way, the participant will be able to achieve true health benefits and reduced risks of co-morbidities due to obesity and the MetS. Comparison with a control group will determine if the treatment is more effective than standard of care for this population.

Motivation and readiness to change:

It is important to assess motivation and readiness to change in individuals who wish to achieve significant life style behavior changes (Ceccarini, M., et al., (2015). Studies have shown that risk of disease development can motivate people to adopt new habits. In a randomized study of weight loss in women at high risk for breast cancer, Hartman, et al (2016) found that women at risk of developing breast cancer were motivated to improve health through weight loss. Using weight loss technology (My Fitness Pal) and phone contact, this intervention resulted in greater weight loss that that of the control group. They concluded that combining technology supported by phone counselling was effective in weight loss as a treatment for women at increased risk for breast cancer. There are no current studies of the effect of motivation on weight loss in people with the metabolic syndrome. However, it is plausible that given the risks of developing diabetes or heart disease, these people may be more motivated to use the app and pursue weight loss to prevent complications of the MetS.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥30 kg/m2;
* fasting glucose ≥ 100mg/dl
* Access to IPhone or Android phone;
* Willing/able to travel to Rockefeller for all study visits;
* Able to speak and understand English;
* Willing to receive weekly phone coaching calls from investigator;
* Willing to monitor and record daily weight and steps in provided notebook.

At least 2 of the following for women:

* waist circumference ≥88 cm;
* Serum triglycerides ≥150mg/dl to ≤ 500mg/dl;
* HDL cholesterol <50mg/dl;
* Hypertension: treated or >130/85 mm/hg untreated during screening

At least 2 of the following for men:

* Waist circumference ≥ 102 cm;
* Serum triglycerides ≥150mg/dl to ≤ 500mg/dl;
* HDL cholesterol <40mg/dl;
* Hypertension: treated or >130/85 mm/hg untreated during screening;

Exclusion Criteria:

* Diabetes except history of gestational diabetes
* HgA1C greater than 6.5% at screening;
* Pregnancy or intent to become pregnant during study participation (women);
* hypo/hyperthyroidism (based on fasting screening labs);
* currently on steroid therapy;
* currently on weight loss medication;
* history of bariatric weight loss surgery;
* currently on statin therapy;
* participation in a formal weight loss program or using another weight loss app;
* any medical, social or psychological condition that, in the opinion of the investigator, would jeopardize the health or well being of the participant or the integrity of the data.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Baseline up to 3 months
  Change in weight measured from baseline to end of study participation (3 months). Weight loss app with compliance is expected to result in 2-3 kg loss.

SECONDARY OUTCOMES:
Retention | Baseline up to 3 months
  Compare the number of drop outs in each group to determine if there is a difference in motivation to lose weight with the app vs standard of care
Change in waist circumference | Baseline up to 3 months
  Weight loss is expected to reduce central obesity
Change in BMI | Baseline up to 3 months
  Weight loss is expected to result in decreased BMI
Change in body composition by Bod Pod | Baseline up to 3 months
  Weight loss is expected to reduce total fat percentage
Change in metabolic parameters | Baseline up to 3 months
  Improvement in metabolic markers: serum glucose, triglycerides, lipids, White Blood Count,erythrocyte sedimentation rate
Change in blood pressure | Baseline up to 3 months
  Reduction in systolic BP
Change in hemoglobin-A1C % | Baseline up to 3 months
  Weight loss and increased activity is expected to reduce Hemoglobin A1C, and indicator of diabetes
Change in motivation to lose weight and adopt healthier lifestyle | Baseline up to 6 months
  URICA motivation questionnaire will monitor motivation at baseline, 3, and 6 months
Change in quality of life by "SF-12v2" questionnaire | Baseline up to 3 months
  Monitor change in perception of quality of life while losing weight

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Walker, NP, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Society of Clinical Oncology. The state of cancer care in America, 2014: a report by the American Society of Clinical Oncology. J Oncol Pract. 2014 Mar;10(2):119-42. doi: 10.1200/JOP.2014.001386. Epub 2014 Mar 10. No abstract available. PMID 24618075
- [Background] Byrne S, Cooper Z, Fairburn C. Weight maintenance and relapse in obesity: a qualitative study. Int J Obes Relat Metab Disord. 2003 Aug;27(8):955-62. doi: 10.1038/sj.ijo.0802305. PMID 12861237
- [Background] Cefalu WT, Bray GA, Home PD, Garvey WT, Klein S, Pi-Sunyer FX, Hu FB, Raz I, Van Gaal L, Wolfe BM, Ryan DH. Advances in the Science, Treatment, and Prevention of the Disease of Obesity: Reflections From a Diabetes Care Editors' Expert Forum. Diabetes Care. 2015 Aug;38(8):1567-82. doi: 10.2337/dc15-1081. PMID 26421334
- [Background] Duncan JM, Janke EA, Kozak AT, Roehrig M, Russell SW, McFadden HG, Demott A, Pictor A, Hedeker D, Spring B. PDA+: A Personal Digital Assistant for Obesity Treatment - an RCT testing the use of technology to enhance weight loss treatment for veterans. BMC Public Health. 2011 Apr 11;11:223. doi: 10.1186/1471-2458-11-223. PMID 21481253
- [Background] Greene J, Sacks R, Piniewski B, Kil D, Hahn JS. The impact of an online social network with wireless monitoring devices on physical activity and weight loss. J Prim Care Community Health. 2013 Jul 1;4(3):189-94. doi: 10.1177/2150131912469546. Epub 2012 Dec 9. PMID 23799706
- [Background] Hruby A, Hu FB. The Epidemiology of Obesity: A Big Picture. Pharmacoeconomics. 2015 Jul;33(7):673-89. doi: 10.1007/s40273-014-0243-x. PMID 25471927
- [Background] Ogden CL, Carroll MD, Fryar CD, Flegal KM. Prevalence of Obesity Among Adults and Youth: United States, 2011-2014. NCHS Data Brief. 2015 Nov;(219):1-8. PMID 26633046
- [Background] Shaw RJ, Bosworth HB, Silva SS, Lipkus IM, Davis LL, Sha RS, Johnson CM. Mobile health messages help sustain recent weight loss. Am J Med. 2013 Nov;126(11):1002-9. doi: 10.1016/j.amjmed.2013.07.001. Epub 2013 Sep 16. PMID 24050486
- [Background] Spring B, Duncan JM, Janke EA, Kozak AT, McFadden HG, DeMott A, Pictor A, Epstein LH, Siddique J, Pellegrini CA, Buscemi J, Hedeker D. Integrating technology into standard weight loss treatment: a randomized controlled trial. JAMA Intern Med. 2013 Jan 28;173(2):105-11. doi: 10.1001/jamainternmed.2013.1221. PMID 23229890
- [Background] DeSilver, Drew. (2016). What's on your table? How America's diet has changed over the decades. Pew Research Center. Retrieved from: http:www.pewresearch.org/fact-tank/2016/12/13/whats-on-your-table-how-americas-diet-has-changed-over-the-decades/
- [Background] American Board of Obesity Medicine. www.abom.org
- [Background] Center for Disease and Prevention (CDC). (2017). Obesity trends among U.S. adults. Retrieved from: www.cdc.gov/obesity/data/prevalence-maps.html
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Background] Ceccarini M, Borrello M, Pietrabissa G, Manzoni GM, Castelnuovo G. Assessing motivation and readiness to change for weight management and control: an in-depth evaluation of three sets of instruments. Front Psychol. 2015 May 11;6:511. doi: 10.3389/fpsyg.2015.00511. eCollection 2015. PMID 26029126
- [Background] Hartman SJ, Nelson SH, Cadmus-Bertram LA, Patterson RE, Parker BA, Pierce JP. Technology- and Phone-Based Weight Loss Intervention: Pilot RCT in Women at Elevated Breast Cancer Risk. Am J Prev Med. 2016 Nov;51(5):714-721. doi: 10.1016/j.amepre.2016.06.024. Epub 2016 Sep 2. PMID 27593420
- See also: Prevalence of the metabolic syndrome in the United States, 2003-2012. — https://www.ncbi.nlm.nih.gov/pubmed/25988468
- See also: DeSilver, Drew (2016) Pew Research Center — http://www.pewresearch.org/fact-tank/2016/12/13/whats-on-your-table-how-americas-diet-has-changed-over-the-decades/
- See also: American Board of Obesity Medicine — http://www.abom.org
- See also: Practical Guide to the Identification, Evaluation, and Treatment of Overweight and Obesity in Adults. National Institutes of Health. National Heart, Lung, and Blood Institute. NIH Publication Number 00-4084. October 2000 — https://www.nhlbi.nih.gov/files/docs/guidelines/prctgd_c.pdf